CLINICAL TRIAL: NCT06597942
Title: Protocol for Maintaining and Improving Mental Status in Alzheimer's Disease (PROMIS-AD): a Pilot Study of Repetitive Transcranial Magnetic Stimulation of the Precuneus for Alzheimer&Amp;Amp;#39;s Disease
Brief Title: Deep Repetitive Transcranial Magnetic Stimulation (rTMS) of the Precuneus for Alzheimer Disease (AD)
Acronym: PROMIS-AD
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Michael K Leuchter, Fellow Physician, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 24-000811
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Alzheimer&Amp;Amp;#39;s Disease; Alzheimer Disease; Dementia Alzheimer Type; Mild Alzheimer&Amp;Amp;#39;s Disease; Moderate Alzheimer&Amp;Amp;#39;s Disease; Alzheimer&Amp;#39;s Disease (AD); Alzheimer&Amp;#39;s Dementia
Keywords: Clinical Trial; deep repetitive transcranial magnetic stimulation (deep rTMS); precuneus; Mild-to-Moderate Probable Alzheimer's Dementia
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: The first stage will involve 5-10 participants receiving open-label active treatment to refine the protocol. After refinement, the second stage will consist of a 1:1 randomized, double-blind, sham controlled clinical trial to study feasibility and tolerability while exploring target engagement and short-term efficacy for memory. Participants will undergo 16 total rTMS brain stimulation sessions over the course of 5 weeks. A full course of open-label active treatment will be offered as an extension to the sham group after unblinding.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Open-Label Active deep rTMS (Experimental): The first stage of the study will consist of protocol refinement. In this first stage of 5-10 participants, all participants will receive open-label active treatment.
  Treatment will consist of 16 sessions of deep rTMS spread over 5 weeks. The induction phase of treatment will be 4 sessions per day for 3 consecutive days (with 60 minutes between sessions), followed by 1 session per week for 4 weeks.
  Individual sessions will consist of 1600 pulses of 20Hz rTMS delivered in 40 pulse trains to the precuneus (using MRI structural neuronavigation) at 100% of depth-corrected motor-threshold with a 28 second intertrain interval (roughly 20 minutes per session).
  Interventions: Device: TMS
- Randomized Active deep precuneus rTMS (Experimental): The second stage of the study will consist of both active and sham treatment groups. Treatment will consist of 16 sessions of deep rTMS spread over 5 weeks. The induction phase of treatment will be 4 sessions per day for 3 consecutive days (with 60 minutes between sessions), followed by 1 session per week for 4 weeks. Individual sessions will consist of 1600 pulses of 20Hz rTMS delivered in 40 pulse trains to the precuneus (using MRI structural neuronavigation) at 100% of depth-corrected motor-threshold with a 28 second intertrain interval (roughly 20 minutes per session). The active group will receive this protocol using an active treatment coil delivering real rTMS.
  Interventions: Device: TMS
- Randomized Sham deep precuneus rTMS (Sham Comparator): The second stage of the study will consist of both active and sham treatment groups. Treatment will consist of 16 sessions of deep rTMS spread over 5 weeks. The induction phase of treatment will be 4 sessions per day for 3 consecutive days (with 60 minutes between sessions), followed by 1 session per week for 4 weeks. Individual sessions will consist of 1600 pulses of 20Hz rTMS delivered in 40 pulse trains to the precuneus (using MRI structural neuronavigation) at 100% of depth-corrected motor-threshold with a 28 second intertrain interval (roughly 20 minutes per session). The placebo group will receive this protocol using a sham TMS coil delivering inactive rTMS.
  Participants in the sham/placebo group will be offered a full open-label extension treatment course of active rTMS on completion of the randomized phase.
  Interventions: Device: TMS; Device: Transcranial Magnetic Stimulation Sham

INTERVENTIONS:
Device: TMS — rTMS Stimulation Parameters Pulse count: 1600 pulses Frequency: 20Hz Pules per train: 40 pulses Inter-train interval: 28 seconds Intensity: 100% Motor Threshold (depth-corrected from MRI) Target: Precuneus using structural MRI navigation with MNI coordinates
  Other Names: precuneus deep repetitive transcranial magnetic stimulation
Device: Transcranial Magnetic Stimulation Sham — Sham coil placed in same location and set with same parameters as active treatment coil. However, this device will not output active treatment and scalp electrodes will mimic the sensation of rTMS for the participant.
  Arms: Randomized Sham deep precuneus rTMS

SUMMARY:
The goal of this clinical trial is to learn if using deep repetitive transcranial magnetic stimulation (rTMS) targeting the precuneus is feasible, tolerable, and potentially efficacious for memory in Probable Alzheimer's Dementia. Previous work studying rTMS in Alzheimer's is mixed, but recent work studying rTMS of the precuneus is encouraging for both its short-term and long-term effects. The main questions this study aims to answer are:

* Is deep rTMS of the precuneus feasible and tolerable in Alzheimer's?
* Are there signs of positive brain changes in response to deep rTMS?
* Is deep rTMS potentially efficacious for memory in Alzheimer's? Researchers will compare active stimulation to placebo stimulation while obtaining memory testing and measurements of the brain (imaging, scalp electrode measurements, bloodwork) to see if active treatment works to treat mild-to-moderate probable Alzheimer's Dementia.

Participants will:

* Engage with memory testing, brain scans, and bloodwork during a comprehensive assessment
* Visit the clinic 3 times for 12 consolidated rTMS sessions, followed by 4 once weekly maintenance sessions
* Be offered a full open-label active treatment course after completing their treatment course if they are initially in the placebo group

DETAILED DESCRIPTION:
This study is designed to examine whether non-invasive electromagnetic stimulation of a specific brain region can help improve memory in the short-term in Alzheimer's Disease (AD). AD is a progressive neurodegenerative disease that affects multiple domains, including cognitive (e.g. memory, executive function), behavioral (e.g. wandering, difficulty controlling impulses, irritability), emotional (e.g. anxiety, depression), and functional (e.g. ability to live independently and complete activities of daily living) domains. It is also associated with increased caregiver burden, which can adversely affect caregivers' health.

One increasingly apparent contributor to disease progression in AD is brain network dysregulation, particularly within the default mode network. Repetitive transcranial magnetic stimulation (rTMS) is a noninvasive therapeutic modality that can be used to stimulate the precuneus, a key node in the default mode network, and maintain signaling function within the default mode network. Previous studies have shown that targeting the precuneus with rTMS may enhance memory in the short term and delay disease progression and functional decline in AD over longer periods. rTMS protocols that have demonstrated promise for treatment delay have first shown short-term impacts on memory, particularly memory of recent and past events.

We will conduct a two-phase trial of rTMS targeting the precuneus in patients with mild to moderate probable AD focused primarily on determining safety and feasibility and secondarily focused on determining short-term efficacy for memory. Participants will be recruited through fliers, social media, print, and web advertising, as well as referrals from other UCLA studies, UCLA clinics, and known community clinics. The first phase will be a handful of subjects (5-10) receiving active treatment only to refine the protocol. After refinement, the second phase will consist of a randomized, double-blind, sham controlled clinical trial with post-blinding crossover examining both safety and short-term efficacy for memory. Participants will be randomized on a 1:1 ratio to either receive precuneus or sham rTMS.

Participants will undergo 16 total rTMS brain stimulation sessions (each session being about 20 minutes) over the course of 5 weeks. The initial induction 3-day intensive course in which rTMS (or sham) will be applied four times daily with 1-hour breaks between treatments will be followed by a 4-week maintenance course in which stimulation will be applied once weekly.

Participants will undergo a range of assessments including brain imaging and oxygenation, genotyping, eye reactivity to light testing, and brain electrical activity measurements to identify changes that occur in the precuneus and its connected regions over time. Participants will also undergo comprehensive neuropsychological (memory and behavioral) testing at baseline and during follow up. Additionally, participants and their caregivers will complete brief weekly check-ins at each treatment during the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 60-100 at the start of the study
* Established diagnosis of Alzheimer's Clinical Syndrome (which is also met through a diagnosis of Alzheimer's Dementia)
* Agreement to participate in study and able to complete informed consent process
* Have a caregiver/study partner who can accompany them to all study visits
* Have a known alternate surrogate decision-maker (in case needed) who can accompany them to the informed consent visit (this person may be the study partner mentioned above)
* Screening MMSE score of 18-26
* Screening GDS score <6
* Either 1) treated with memory-enhancing medication (cholinesterase inhibitor) for at least 2 months, 2) failed trial with no plan to re-trial, or 3) no trial planned during the course of the study for other reasons
* No change in use of psychotropic medication for the treatment of depression, anxiety, ADHD, or psychosis for 2 weeks prior to the study

Exclusion Criteria:

* Participant and/or their surrogate are unwilling or unable to provide informed consent
* Currently pregnant or potentially pregnant
* Diagnosis of a dementia or cognitive disorder due to a cause other than Alzheimer's Disease
* Diagnosis of severe Dementia (CDR > 2.0) at the start of the study
* History of substance use disorder currently not in sustained remission
* Substance misuse within the past 6 months (excluding nicotine or caffeine)
* History of stroke, traumatic brain injury with loss of consciousness, or other major neurologic disorder (e.g., epilepsy, Huntington's disease, Parkinson's disease)
* History of seizure disorder or family history of seizure disorder in a first-degree relative
* Poorly-controlled hypertension, cardiovascular disease, or cerebrovascular disease
* History of any other major active medical, neurologic, or psychiatric illness affecting cognition (associated with cognitive impairment) or a participant's ability to safely and meaningfully participate in the study
* Non-fluent in English (not native or functionally-native)
* Contraindication to TMS or MRI including claustrophobia, MRI-incompatible or unknown metal in body (including facial tattoos with uknown or metallic inks), surgery within 60 days, certain implants (excluding dental fillings), or previous abnormal MRI results.
* Has previous history of TMS treatment in the past (not TMS naïve)
* Currently enrolled in a memory-enhancement study
* Alteration in cognitive-enhancement medication dose within the past 2 months or active plans for dose alteration during the course of the study (previously unplanned changes that occur during the study will be examined on a case-by-case basis)
* History of treatment with lecanemab, aducanumab, donanemab, or other monoclonal antibody treatment for Alzheimer's Disease (due to lack of knowledge surrounding the impacts of these treatments)
* Currently or within the past 2 weeks taking any of the following classes of medication:

  * Anticholinergic (e.g., tolterodine, benztropine)
  * Sedating antihistamines (e.g., diphenhydramine)
  * any drug that has significant anticholinergic or antihistaminic side effects (e.g., tricyclic antidepressant medications, mirtazapine).
  * Benzodiazepines. While not a strict rule out, this will be decided on a case-by-case basis
  * Antiepileptic agents. While not a strict rule out, this will be decided on a case-by-case basis
  * Antipsychotic agents. While not a strict rule out, this will be decided on a case-by-case basis

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-10-17 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Completion Rate | From enrollment to the end of treatment after 5 weeks
  The percentage/fraction of participants who complete the full course of study treatment

SECONDARY OUTCOMES:
Adverse Events | From enrollment until the end of treatment at 5 weeks
  The incidence of adverse events/side effects during the course of study treatment. Known common side effects of rTMS for other indications include discomfort/pain at the site of stimulation and mild transient headaches. Known rare though serious side effects include seizure (generally 1 in 30,000)
Gray Matter Volume | From pre-treatment baseline structural MRI to post-treatment structural MRI
  There are indications rTMS may preserve gray matter volume in neurodegenerative disease near the site of stimulation and connected areas. Volume of the precuneus, stimulated areas, and connected areas will be studied before and after treatment.
EEG | From pre-treatment EEG to post-treatment EEG after 5 weeks
  Beta and Gamma Oscillatory power, as well as Beta/Theta periodic power ratios will be examined.
NIH Cognitive Toolbox | Enrollment to end of 5 weeks of treatment
  The NIH Cognitive Toolbox consists of a battery of tests well-validated for memory testing. Participants will undergo testing with this tool before and after completing treatment.
resting-state functional MRI connectivity | from enrollment to the end of treatment at 5 weeks
  Participants will undergo resting-state functional blood-oxygen-level dependent (BOLD) MRI (rs-fMRI) to examine functional connectivity between the precuneus and other areas of the brain, particularly within the default mode network
Repeatable Battery for the Assessment of Neuropsychological Status Update (RBANS Update) | From pre-treatment to post-induction pre-maintenance to end-of-treatment after 5 weeks.
  The RBANS Update is a well-established neuropsychological test for memory. Participants will undergo testing with the RBANS before treatment, between induction and maintenance treatment, and after completing treatment. Scores range from 40 to 160, with higher scores indicating better performance and lower scores indicating worse performance.
Clinical Dementia Rating Scale (CDR) | From enrollment to the end of treatment at 5 weeks
  CDR score and CDR-SB (sum of boxes score) are gathered from the CDR, an interview-based measure of global dementia severity. Participants and caregivers engage in interview. Global scores range from 0 to 3 with higher scores indicating greater severity of dementia. Sum of boxes scores range from 0 to 18 with higher scores indicating greater severity of dementia.

OTHER OUTCOMES:
Zarit Burden Index | From enrollment to end of treatment at 5 weeks
  The caregiver(s) of participants will complete this self-report measure of caregiver burden, with multiple versions available. It is one of the most widely-used and validated assessments of caregiver burden
Neuropsychiatric Inventory (NPI) | From enrollment to the end of treatment at 5 weeks
  Participants and caregivers engage in comprehensive interview to assess the presence and severity of ten behavioral and two neurovegetative symptoms common in AD. This will aid in assessment of behavioral and emotional domains
ADL/IADL | From enrollment to the end of treatment at 5 weeks
  Participants and caregivers engage in a discussion of participant's ability to complete and/or level of assistance needed to complete everyday tasks. This will aid in assessment of everyday function and overall dependence on others.
Peripheral Tau and Amyloid levels | from enrollment to end of treatment at 5 weeks
  Participants will undergo a blood draw for the purpose of determining peripheral Tau and Amyloid burden as a potential marker of AD pathology and allow researchers to explore potential changes with treatment.
Pupillary Reactivity | from enrollment to the end of treatment at 5 weeks
  Participants will undergo measurement of their pupillary light response using a brief flash of light.
Geriatric Depression Scale (GDS) | From enrollment to the end of treatment at 5 weeks
  Participants will complete this self-report depression rating scale; it is a self-report rating scale designed and validated in older populations for late life depression. Scores range from 0 to 30, with higher scores indicating a greater depressive symptom burden.
Neuropsychiatric Inventory--Questionnaire | From enrollment to the end of treatment at 5 weeks
  This is the abbreviated self-report version of the NPI. Though it is not as comprehensive as the NPI, it is useful as a tool tracking in a longitudinal fashion due to its briefer nature. The NPI-Q generates two scores, a severity score (range 0-36) and a frequency score (0-60); higher scores indicate greater burden/level of impairment/worse outcome.
Mini-Mental State Examination (MMSE) | from enrollment to the end of treatment at 5 weeks
  Participants engage in a structured brief memory assessment lasting approximately 15 minutes. Scores range from 0-30, with higher scores indicating better performance/outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Leuchter, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA TMS Clinical and Research Service, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Demographics, neuropsychological outcomes, pupillary reactivity, blinding validation, tau and amyloid levels, APOE status, EEG, MRI.
  EEG and imaging data may not include raw EEG or imaging data, but will likely instead consist of data extracted from EEGs and MRIs.
Supporting Information: SAP
Time Frame: Beginning within 12 months of publishing results and ending no sooner than 3 years after publication of results.
Access Criteria: After completion of the study, de-identified data may be made available to other institutions or secure online databases on reasonable request (such as Clinical Study Data Request, https://www.clinicalstudydatarequest.com). All other data will be handled the same way it is handled during the study.

REFERENCES:
- [Derived] Leuchter MK, Oughli HA, Durbin KA, Jackson NJ, Elashoff D, Chang TS, Corlier J, Ngo D, Matthews C, Wong D, Fogel BL, Bitan G, Leuchter AF, Vossel K, Suthana N. Broad repetitive transcranial magnetic stimulation (rTMS) of the precuneus in Alzheimer's disease: A rationale and study design. Alzheimers Dement (N Y). 2025 Mar 10;11(1):e70043. doi: 10.1002/trc2.70043. eCollection 2025 Jan-Mar. PMID 40065917